CLINICAL TRIAL: NCT06626984
Title: Investigation of Novel and Established Therapies in a Human Intravenous Lipopolysaccharide Model of Sepsis
Acronym: INITIALISE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Medical Research Council (Other Government); The Royal College of Anaesthetists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 22064JS-AS
Record Dates: First submitted 2023-05-03; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Fluid Overload; Endothelial Dysfunction; Microcirculation
Keywords: Intravenous Fluid Therapy; Imatinib
MeSH Terms: conditions — Sepsis; Edema | interventions — Imatinib Mesylate; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: The first 5 participants recruited to this study will receive intravenous fluid therapy only. This will allow us to directly elucidate the effects of intravenous fluid therapy on markers of vascular injury, markers of systemic inflammation, microcirculatory function and venous congestion in healthy volunteers.
  After the first 5 participants have completed the interventions, a 2x2 factorial design will be adopted, in which participants are randomised to:
  1. Intravenous fluids or no intravenous fluids, AND TO
  2. Imatinib or no imatinib
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators taking blood samples and performing ultrasound based imaging techniques will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intravenous LPS only (No Intervention): LPS dose 2ng/kg.
- Intravenous LPS AND Intravenous Fluid Therapy* (Experimental): *The first 5 participants recruited to this study will receive intravenous fluid therapy only. This will allow us to directly elucidate the effects of intravenous fluid therapy on markers of vascular injury, markers of systemic inflammation, microcirculatory function and venous congestion in healthy volunteers.
  LPS dose 2ng/kg. Intravenous fluid 30ml/kg in total (maximum volume of 2500mls). Administered in two divided doses (15mls/kg) intravenously. Each bolus will be administered at a fixed rate of 999mls/hr. The administration is to commence 90 minutes following intravenous LPS.
  Interventions: Drug: Compound sodium lactate solution
- Intravenous LPS AND Imatinib Therapy (Experimental): LPS dose 2ng/kg. Imatinib 600mg 1 hour prior to LPS administration.
  Interventions: Drug: Imatinib
- Intravenous LPS AND Intravenous Fluid Therapy AND Imatinib Therapy (Experimental): LPS dose 2ng/kg. Intravenous fluid 30ml/kg in total (maximum volume of 2500mls). Administered in two divided doses (15mls/kg) intravenously. Each bolus will be administered at a fixed rate of 999mls/hr. The administration is to commence 90 minutes following intravenous LPS.
  Imatinib 600mg 1 hour prior to LPS administration.
  Interventions: Drug: Imatinib; Drug: Compound sodium lactate solution

INTERVENTIONS:
Drug: Imatinib — Pre-treatment with 600mg Imatinib administered 1 hour prior to intravenous LPS.
  Arms: Intravenous LPS AND Imatinib Therapy; Intravenous LPS AND Intravenous Fluid Therapy AND Imatinib Therapy
Drug: Compound sodium lactate solution — Total of 30 ml/kg administered 90 minutes following intravenous LPS. 30mls/kg (maximum volume of 2500mls) administered in two divided doses (15mls/kg) intravenously. Each bolus will be administered at a fixed rate of 999mls/hr.
  Arms: Intravenous LPS AND Intravenous Fluid Therapy AND Imatinib Therapy; Intravenous LPS AND Intravenous Fluid Therapy*

SUMMARY:
Sepsis is a common and life-threatening condition caused by a dysregulated host immune response to infection. Given the prominent role of endothelial breakdown and dysfunction in sepsis, therefore, there is an urgent need to establish strategies to protect the endothelium and preserve microcirculatory function.

This study is a randomised clinical study investigating intravenous fluid therapy and oral imatinib therapy in healthy human volunteers exposed to intravenous lipopolysaccharide (LPS).

The objective of the study is to investigate the biological effects of fluid and imatinib therapy on LPS-induced microcirculatory dysfunction.

DETAILED DESCRIPTION:
The benefits of intravenous fluid administration in sepsis remain uncertain. A growing body of evidence suggests that excessive fluid administration is harmful. An association between a more positive fluid balance and mortality in critically ill patients has been repeatedly demonstrated. Moreover, emerging evidence suggests that intravenous fluid administration induces glycocalyx injury, thought to be mediated by shear stress. In sepsis the rapid administration of intravenous fluids is hypothesised to exacerbate glycocalyx injury, capillary leak and tissue oedema formation.

Recent work has highlighted the protective effects of Imatinib, a tyrosine kinase inhibitor, on endothelial barrier function in animal models of microcirculatory dysfunction as well as in patients with endothelial barrier dysfunction. Moreover, Imatinib has also been demonstrated to attenuate markers of systemic inflammation in animals with a LPS-induced lung injury model of acute respiratory distress syndrome. There is, therefore, a growing body of evidence to support a potential therapeutic role for Imatinib in disease states involving inflammatory vascular leak.

The hypothesis being tested is that:

1. Intravenous fluid therapy will exacerbate the degree of vascular dysfunction and systemic inflammation observed in this model.
2. Imatinib pre-treatment will attenuate the degree of vascular dysfunction and systemic inflammation observed in this model.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged between 18 and 40 years of age
2. Informed consent to participate

Exclusion Criteria:

1. Current participation in a clinical trial
2. Pregnant or breastfeeding
3. Current history of smoking
4. Alcohol intake > 21 units per week
5. Regular intake of any relevant prescription or over-the-counter medication. Any regular medication use will be reviewed on a case-by-case basis as to (a) risk and (b) potential confounding effect.
6. Oxygen saturation <95% breathing room air
7. Abnormal findings on history, examination or laboratory tests suggestive of underlying illness (in the opinion of the clinician undertaking screening)
8. History of recurrent vaso-vagal episodes
9. Allergy to Imatinib
10. Positive or equivocal hepatitis B or C serology result

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of vascular and glycocalyx injury | Up to 8 hours following LPS administration
  Change in plasma biomarkers of vascular and glycocalyx injury including but not limited to - Hyaluronan

SECONDARY OUTCOMES:
Biomarkers of inflammation | Up to 8 hours following LPS administration
  Change in plasma biomarkers of inflammation including but not limited to - Interleukin-6
Venous Excess Ultrasound Score | Up to 8 hours following LPS administration
  Ultrasound measure of venous congestion
B-lines | Up to 8 hours following LPS administration
  Ultrasound measure of pulmonary oedema

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available to share with other researchers. Anonymised data will be grouped into a database which may be shared with other researchers.